CLINICAL TRIAL: NCT00206856
Title: Rapid Assessment of Bedside BNP In Treatment of Heart Failure (RABBIT)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Abbott RDx Cardiometabolic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 001
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Triage® B-Type Natriuretic Peptide (BNP) Test

SUMMARY:
To determine the clinical utility of using the Triage® BNP Test to guide therapy in outpatients with heart failure

DETAILED DESCRIPTION:
The Triage® BNP Test has been cleared by the U.S. Food and Drug Administration as an aid in the diagnosis and assessment of severity of heart failure. In addition to numerous reports describing the diagnostic and prognostic utility of BNP, reports from various pilot studies have described decreases in BNP in association with various heart failure therapies. Other reports have described modest increases in BNP in association with digitalis and beta-receptor antagonism. The observation that the circulating BNP concentration decreases during heart failure therapy, coupled with the ability of BNP to be used as a prognostic tool and assess the severity of heart failure, it is hypothesized that using BNP measurements to guide heart failure therapy could have a significant impact on the care of heart failure patients. This hypothesis is supported by various reports of pilot studies that describe a significant benefit of administering therapy tailored to concentrations of BNP and related peptides. Patients that are discharged after a hospitalization for heart failure will be approached for study enrollment.This is a multi-center, single (patient)-blinded cluster-randomized study. Half of the sites will have BNP measurements available to guide therapy (experimental arm) and the other half of the sites will not have BNP measurements available (control arm). Blood (plasma) will be collected at each visit and appropriate forms completed. Patients will be asked to complete a Minnesota living with heart failure questionnaire and to do a 6-minute walk test. Patients will be followed for 12 months.

ELIGIBILITY:
Inclusion Criteria:

Age 18 or older Patient was hospitalized and treated for heart failure Patient is fully stabilized at discharge Able to give informed consent

Exclusion Criteria:

History of severe pulmonary disease Chronic O2 therapy for COPD Primary pulmonary hypertension History of renal disease requiring dialysis History of severe hepatic disease Patients using LVAD's Stroke, MI, PTCA, CABG or unstable angina within the past 1 month Bi-ventricular pacemaker placement within last 1 month History of severe aortic stenosis History of severe mitral stenosis History of constrictive pericarditis Patient has had a cardiac transplant Status 1 cardiac transplant candidates ICD or DRG assignment of non-Q wave MI within last 1 month Patient has cor pulmonale A re-hospitalization, death or an IV treatment for heart failure before the first post-discharge visit and/or15) Planned chronic IV treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720
Dates: Start 2003-07; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Combined endpoint of mortality, unplanned clinic or hospital visits that require IV treatment for heart failure, and quality of life.

SECONDARY OUTCOMES:
All-cause re-hospitalization, Quality of Life, 6 minute walk distance, New York Heart Association class and BNP.

CONTACTS AND LOCATIONS:
Overall Officials: James B Young, MD, Principal Investigator — The Cleveland Clinic
Locations (29):
- United States (29):
  - Scottsdale CardiovascularResearch, Scottsdale, Arizona
  - San Diego Veterans Administration Hospital, San Diego, California
  - San Francisco Veterans Administration Hospital, San Francisco, California
  - Denver Veterans Administration Hospital, Denver, Colorado
  - Cardiology Associates of Fort Lauderdale, Fort Lauderdale, Florida
  - Shands at the University of Florida, Gainsville, Florida
  - VNH Heart Center Research, Port Charlotte, Florida
  - Heart and Vascular Institute of Florida, St. Petersburg, Florida
  - Northwestern University Memorial, Chicago, Illinois
  - Midwest Heart Institute, Lombard, Illinois
  - Advocate Health, Oak Lawn, Illinois
  - Oschner Clinic, New Orleans, Louisiana
  - University Mass. Memorial Hospital, Worcester, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - William Beaumont Hospital-Troy, Troy, Michigan
  - Minnesota Veterans Administration, Minneapolis, Minnesota
  - Medicor Cardiology, Bridgewater, New Jersey
  - Buffalo Heart Group,, Buffalo, New York
  - Cardiovascular Medical Associates, Garden City, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - South Bay Cardiovascular Associates, West Islip, New York
  - Carolinas Medical Center/Sanger Clinic, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Cleveland University Hospital, Cleveland, Ohio
  - Baylor College of Medicine, Houston, Texas
  - San Antonio VA Medical Center, San Antonio, Texas
  - Latter Day Saints Hospital, Salt Lake City, Utah